CLINICAL TRIAL: NCT01866696
Title: Computer Assisted Implant Surgery and Immediate Loading With Full-arch Screw Retained Prosthesis
Brief Title: Computer Assisted Implant Surgery and Immediate Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Clinical Professor, Università degli Studi di Sassari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID051313
Record Dates: First submitted 2013-05-13; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Edentulous Jaws
Keywords: Computer assisted implant surgery,; Immediate loading,; CAD/CAM
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- guided implant insertion and immediate loading (Experimental): This work was designed as a prospective case series clinical study. Twenty patients have been consecutively rehabilitated with an immediately loaded oral implant supported fixed full prosthesis. A total of 120 oral implants (Nobel Replace Tapered Groovy; Nobel Biocare AB, Goteborg, Sweden) supporting 23 bridges (8 mandible, 15 maxilla) were placed , 22 of which in fresh post extraction sockets. 117 out of 120 oral implants were immediately loaded.
  Interventions: Device: oral implants

INTERVENTIONS:
Device: oral implants — For all cases, the following surgical and prosthetic protocol was followed.:
  * Clinical examination
  * Radiological examination
  * Guided oral implants insertion
  * Immediate Prosthetic loading
  * Follow-up
  Other Names: Oral implants Nobel Replace Tapered Groovy; Nobel Biocare AB, Goteborg, Sweden

SUMMARY:
Purpose: The aim of this study was to analyze the clinical and radiographic outcomes of 23 edentulous jaws treated with 3D software planning, guided surgery, immediate loading and restored with Cad-Cam Zirconia and titanium full arch frameworks.

Material & methods: This study was designed as a prospective clinical trial. Twenty patients have been consecutively rehabilitated with an immediately loaded implant supported fixed full prosthesis. A total of 120 fixtures supporting 23 bridges (8 mandible, 15 maxilla) were placed , 22 of which in fresh post extraction sockets. All the implants were inserted with an insertion torque of 35/45 Ncm. 117 out of 120 implants were immediately loaded the other 3 were delayed loaded.

Outcome measures were implants survival, radiographic marginal bone-levels and bone remodeling, soft tissue parameters and complications.

ELIGIBILITY:
Inclusion criteria were:

-edentulous patients or patients with hopeless teeth in need to be restored with full arches prosthesis

Exclusion criteria were:

* presence of systemic diseases (i.e. haematologic disease, uncontrolled diabetes, serious coagulopathies and diseases of the immune system)
* irradiation to the head or neck region within 12 months before surgery
* presence severe bruxism or clenching habits
* pregnancy
* poor oral hygiene
* poor motivation to return for scheduled follow-up visit

Ages: 39 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
implants survival | 0-30 months

SECONDARY OUTCOMES:
peri-implant bone | 12-30 months
  marginal bone remodeling and marginal bone level

OTHER OUTCOMES:
peri-implant mucosal response | 12-30 months
prosthetic success | 0-30 months
biological and prosthetic complication | 12-30 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvio M Meloni, DDS, Study Director — Università degli Studi di Sassari
Locations (1):
- University of Sassari, Sassari, SS, Italy

REFERENCES:
- [Derived] Meloni SM, De Riu G, Pisano M, Lolli FM, Deledda A, Campus G, Tullio A. Implant Restoration of Edentulous Jaws with 3D Software Planning, Guided Surgery, Immediate Loading, and CAD-CAM Full Arch Frameworks. Int J Dent. 2013;2013:683423. doi: 10.1155/2013/683423. Epub 2013 Jul 29. PMID 23983690